CLINICAL TRIAL: NCT06510543
Title: Goal-directed Enteral Nutritional Therapy for Malnourished Esophageal Cancer Patients During Perioperative Management
Brief Title: Goal-directed Enteral Nutritional Perioperative Management
Acronym: GENTLEMAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, YIN LI, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GENTLEMAN
Record Dates: First submitted 2024-06-18; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Esophagus Cancer
Keywords: Esophageal Cancer; Esophagectomy; Nutritional Therapy; Morbidity; Survival; Malnourished
MeSH Terms: conditions — Esophageal Neoplasms; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal-directed enteral nutritional therapy (Experimental): The participants will be administered a supervised goal-directed nutritional therapy. The enteral nutrition (EN) regimens include homemade meals with or without ORAL IMPACT® according to the daily goal.
  Interventions: Dietary Supplement: Goal-directed EN therapy
- Conventional enteral nutritional therapy (Active Comparator): The participants will be administered with an unsupervised and liberal nutritional support. The EN regimens will not include ORAL IMPACT®.
  Interventions: Dietary Supplement: Conventional EN therapy

INTERVENTIONS:
Dietary Supplement: Goal-directed EN therapy — The participants will be administered a supervised goal-directed nutritional therapy. The enteral nutrition (EN) regimens include homemade meals with or without ORAL IMPACT® according to the daily goal.
  Arms: Goal-directed enteral nutritional therapy
Dietary Supplement: Conventional EN therapy — The participants will be administered the conventional nutritional therapy according to the Chinese expert consensus on perioperative nutritional support in enhanced recovery after surgery (2019 edition).
  Arms: Conventional enteral nutritional therapy

SUMMARY:
This clinical trial aims to determine whether perioperative goal-directed nutritional therapy can prevent postoperative pulmonary and other major complications in malnourished esophageal squamous cell cancer patients. Its main question is whether individualized nutritional therapy can improve short-term surgical outcomes and long-term prognosis. Researchers will compare goal-directed and conventional nutritional therapy to identify differences in morbidities and survival.

DETAILED DESCRIPTION:
Severe malnutrition is a significant risk factor for postoperative complications in esophageal cancer patients. Early oral nutritional supplementation after surgery can prevent weight loss and improve quality of life. The EFFORT trial showed that individual-based enteral nutrition support reduced complications, extended 1-year survival, and improved quality of life. This study aims to assess the safety and effectiveness of individualized perioperative nutrition support guided by daily energy targets in esophageal cancer patients at nutritional risk. It also seeks to determine if supplementing immunonutrition can effectively reduce postoperative complications. This study was conducted as a multicenter, open-label, randomized, controlled phase 3 trial. The experiment group was administered goal-directed enteral nutritional therapy, while the control group received conventional enteral nutritional therapy. The study observed the participants' major pulmonary and other complications within 90 days post-surgery and nutritional status, disease-free survival (DFS), and overall survival (OS) in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years old;
2. ECOG PS 0~1;
3. NRS 2002 score ≥3;
4. Malnutrition diagnosed according to the GLIM criteria;
5. Histopathologically confirmed as esophageal squamous cell carcinoma;
6. Primary tumors located in thoracic esophagus;
7. Resectable locally advanced disease with clinical stage II to IVA (8th edition UICC/AJCC) evaluated by a multidisciplinary team;
8. Neoadjuvant therapy will be administered, which may entail preoperative chemo-radiotherapy, chemotherapy only, or a combination of immunotherapy such as anti-PD-1/PD-L1;
9. Informed consent for random assignment and completion of the protocol.

Exclusion Criteria:

1. NRS 2002 score < 3;
2. Upfront surgery without neoadjuvant treatment;
3. Any comorbidity interferes with the digestion and absorption of ORAL IMPACT®;
4. Receiving any other nutritional support during the study;
5. Unable to consume nutrition orally or receive it through tube feeding before surgery;
6. History of other malignancies in the past 5 years, except successfully treated basal-cell skin carcinoma and cervical tumors in situ;
7. Severe abnormalities of liver and kidney functions (ALT≥2 times the upper limit of normal; Total bilirubin Tbil≥2 upper limit of normal; Creatinine Cr≥2 upper limit of normal);
8. Metabolic disorders, including uncontrolled diabetes mellitus or fasting blood glucose ≥10mmol/L, hypothyroidism, or hyperthyroidism;
9. Receiving fat emulsion containing Omega-3 fatty acids, glutamine, thymosin, glucocorticoid, thyroxine, growth hormone, and anti-tumor necrosis factor biologic agents
10. History of known allergy to any component of ORAL IMPACT®;
11. Pregnant or lactating women, women of childbearing potential with either a positive pregnancy test at baseline or not using a reliable and appropriate contraceptive method;
12. Refuse to sign the consent or unable to follow the study protocol;
13. Inappropriate to participate in this study judged by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2031-05-30 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative pulmonary complications | Randomization to three months after surgery
  According to the Esophagectomy Complications Consensus Group (ECCG) standardization of complications reporting, pulmonary complications include pneumonia, pleural effusion, pneumothorax, atelectasis, mucous plugging, respiratory failure, acute respiratory distress syndrome, acute aspiration, tracheobronchial injury, and prolonged air-leak.
Rate of unplanned hospital admissions | Randomization to three months after surgery
  Any admission (all cause) for an unforeseen or unplanned (non-elective) cause within 90 days of discharge from an index acute hospital admission.
Rate of unplanned ICU admission | Randomization to three months after surgery
  Any admission (all cause) for an unforeseen or unplanned (non-elective) cause within 90 days of discharge from an index acute ICU admission.
Overall survival | Randomization to five years
  The time from randomization to death. Any patients lost to follow up or still alive at the time of evaluation are censored.

SECONDARY OUTCOMES:
Rate of postoperative non-pulmonary complications | Randomization to three months after surgery
  Non-pulmonary complications according to the ECCG standardization of complications reporting.
Level of serum prealbumin | Randomization to three months after surgery
  Prealbumin, also known as transthyretin, has a half-life in plasma of ∼2 days, much shorter than that of albumin. Prealbumin is therefore more sensitive to changes in protein-energy status than albumin, and its concentration closely reflects recent dietary intake rather than overall nutritional status.
Body mass index (BMI) | Randomization to three months after surgery
  A person's weight in kilograms divided by the square of height in meters.
Lean body mass | Randomization to three months after surgery
  The weight of the body minus the⁣ fat content, representing the amount of⁣ muscle, bone, and organs in the body.
Rate of treatment-related adverse events (TRAEs) | Randomization to three months after surgery
  An event that emerges during treatment having been absent pre-treatment, or worsens relative to the pre-treatment state.
Rate of R0 resection | Randomization to three months after surgery
  Distance between tumor and the circumferential resection margin (CRM) more than 1 mm.
Rate of pathologic complete response (pCR) | Randomization to three months after surgery
  The absence of invasive/in situ cancer in the resected esophagus and regional lymph nodes.
Disease-free survival (DFS) | Randomization to five years
  Defined as the proportion of patients without disease progression or death.
Scale of health-related quality of life (HRQOL) | Randomization to three months after surgery
  A state of complete physical, mental and social well-being, and not merely the absence of disease and infirmity evaluated by EORTC OES18、EQ-5D、FAACT.

CONTACTS AND LOCATIONS:
Overall Officials: Yin Li, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (17):
- China (17):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Daping Hospital, Third Affiliated Hospital of Third Military Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Anyang Cancer Hospital, Anyang, Henan
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Changzhi People's Hospital, Changzhi, Shanxi
  - Shanxi Cancer Hospital, Chinese Academy of Medical Sciences, Taiyuan, Shanxi
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No